CLINICAL TRIAL: NCT00857480
Title: A Single-Centre, Open, Controlled, Randomised Cross-Over Study in Healthy Male and Female Volunteers to Evaluate the Pharmacokinetics of Cholyl-Lysyl-Fluorescein (NRL972) in the Presence of Medication-Induced Changes in Cytochrome P450 or Biliary Transporter Proteins. Part B: Interaction With Ursodeoxycholic Acid and Cloxacillin
Brief Title: Evaluation of the PK of NRL972 Following Pre- and co-Administration of Ursodeoxycholic Acid and Cloxacillin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-05/2005 (IN-B)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference (Experimental): No pre-treatment
  Interventions: Drug: NRL972
- T1 (Experimental): Cloxacillin pre- and co-treatment
  Interventions: Drug: NRL972
- T2 (Experimental): UDCA pre-treatment
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — Single intravenous administration of 2 mg NRL972
  Arms: Reference
Drug: NRL972 — Pre-treatment and co-treatment with 1 g Cloxacillin t.i.d. for three days from the morning of D-3 until the morning of Day D01 0:30 hour before the intravenous administration of NRL972.
  Arms: T1
Drug: NRL972 — Three week pre-treatment with daily doses of 500 mg b.i.d ursodeoxycholic acid from the morning of D-20 until the evening of Day D-1
  Arms: T2

SUMMARY:
A study in healthy volunteers to determine whether different drugs metabolised by the liver have any effects on how NRL972 is processed within the body.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females (females of non-childbearing potential or of childbearing potential while taking medically appropriate contraception)
2. Caucasian
3. Age: 21 - 40 years
4. BW 50 - 100 kg
5. BMI 20 - 26 kg.m-2
6. healthy based on the pre-study examination
7. willing and able to provide informed consent

Exclusion Criteria:

General - all subjects

1. Previous participation in the trial
2. Participant in any other trial during the last 90 days
3. Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months
4. History of any clinically relevant allergy (including hypersensitivity to the trial medications)
5. Presence of acute or chronic infection
6. Presence or history of any relevant co-morbidity
7. Resting systolic blood pressure > 160 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
8. Clinically relevant ECG-abnormalities, prolonged QTc with > 450 msec in males and > 460 msec in females in particular
9. Presence of any relevant abnormality in the laboratory safety tests, especially low haemoglobin, increased liver enzymes
10. Positive serology for HBsAg, anti HBc and anti HCV
11. Positive HIV test
12. Positive alcohol or urine drug test on recruitment (and upon admission)
13. History of alcohol and/or drug abuse and/or daily use of > 30 gr alcohol
14. Smoking more than 15 cigarettes/day or equivalent of other tobacco products
15. Use of prohibited medication
16. Suspicion or evidence that the subject is not trustworthy and reliable
17. Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard

    General - all females
18. Positive pregnancy test
19. Lactating
20. Not using appropriate contraception in pre-menopausal women (note: under the conditions of the present study, women using hormonal contraceptives will be informed that this method is not sufficient during the study and that further i.e. mechanical methods [condom, diaphragm with spermicidal gel] should be us

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Total clearance by non-compartmental analysis. Apparent terminal disposition half-life t½ by non-compartmental analysis | 4 hours post-dose

SECONDARY OUTCOMES:
Non-compartmental PK-analysis based on the extensive profile (up to last quantifiable data point), the 'short' profile (over the first hour after injection), and the two-point profile based on selected data-pairs over the 1st hour after dosing | 4 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; Emil Gatchev, PD Dr med, Principal Investigator — MHAPT "Zarita Johanna" University Hospital
Locations (1):
- MHAPT "Zarita Johanna" University Hospital, Sofia, Bulgaria